CLINICAL TRIAL: NCT00843492
Title: A Multicentre, Randomized, Open-label Study to Evaluate the Efficacy andSafety of Fondaparinux Versus Low Molecular Weight Heparin(Nadroparin) in Patients Requiring Rigid or Semi-rigid Immobilization for at Least 21 Days and up to 45 Days Because of Isolated Non-surgical Below-Knee Injury
Brief Title: A Study to Evaluate the Efficacy and Safety of Fondaparinux for the Prevention of Venous Blood Clots in Patients With a Plaster Cast or Other Type of Immobilization for a Below-knee Injury Not Needing Surgery
Acronym: FONDACAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109350
Record Dates: First submitted 2008-12-11; First posted 2009-02-13 (Estimated); Results first posted 2012-07-18 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2014-02

CONDITIONS: Thrombosis, Venous
Keywords: deep vein thrombosis; immobilization; nadroparin; isolated lower-extremity injuries distal to the knee; plaster cast; non-surgical leg injury; venous thromboembolism; bleeding events; fondaparinux
MeSH Terms: conditions — Venous Thrombosis; Venous Thromboembolism | interventions — Fondaparinux; Nadroparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nadroparin (Active Comparator): After randomization (Day 1), subjects will receive subcutaneously once daily nadroparin 2850 anti-Xa IU (0.3 mL) for at least 21 Days, up to complete mobilization, corresponding to cast or brace removal. The maximal duration of treatment is 45 days. Patients will then be followed up to five weeks (± one week) after the cast or brace removal.
  Interventions: Drug: Nadroparin
- Fondaparinux (Experimental): After randomization (Day 1), subjects will receive subcutaneously, once daily, fondaparinux 2.5 mg (1.5 mg in patients with creatinine clearance between 30 and 50 mL/min) for at least 21 Days, up to complete mobilization, corresponding to cast or brace removal. The maximal duration of treatment is 45 days. Patients will then be followed up to five weeks (± one week) after the cast or brace removal.
  Interventions: Drug: Fondaparinux sodium

INTERVENTIONS:
Drug: Fondaparinux sodium — After randomization (Day 1), subjects will receive subcutaneously once daily fondaparinux 2.5 mg [0.5mL] (1.5 mg [0.3mL] in patients with creatinine clearance between 30 and 50 mL/min) for at least 21 Days, up to complete mobilization, corresponding to cast or brace removal. The maximal duration of treatment is 45 days.
  Arms: Fondaparinux
Drug: Nadroparin — After randomization (Day 1), subjects will receive subcutaneously once daily nadroparin 2850 anti-Xa IU (0.3 mL) for at least 21 Days, up to complete mobilization, corresponding to cast or brace removal. The maximal duration of treatment is 45 days.
  Arms: Nadroparin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of fondaparinux in comparison with a heparin (nadroparin) in preventing deep vein thrombosis (blood clots in the leg veins), whether symptomatic or detected by ultrasound, and pulmonary embolism (blood clots that migrate to the lungs) in patients with leg injuries below the knee that require a cast or other type of immobilization but not surgery.

DETAILED DESCRIPTION:
The study is designed to evaluate the efficacy and safety of fondaparinux sodium 2.5 mg (1.5 mg in patients with a creatinine clearance between 30 and 50 mL/min) once daily versus Low-Molecular Weight Heparin (nadroparin 2850 anti-Xa IU, 0.3 mL, once daily), with respect to the occurrence of venous thromboembolism, death and bleeding complications in patients requiring rigid or semi-rigid immobilization for at least 21 days and up to 45 days because of isolated nonsurgical below-knee injury. Treatment will be continued up to complete mobilization, e.g. plaster cast or brace removal, for a maximum of 45 days. The study will be a European, multicentre, randomized, open-label, controlled, two-parallel-group, phase III study in 1350 male and female patients 18 years of age or older, presenting with at least one additional major risk factor for VTE. After randomization (Day 1), subjects will receive subcutaneously, once daily, either fondaparinux or nadroparin up to complete mobilization. After cast or brace removal, a systematic, bilateral compression ultrasound will be done in all patients. Patients will be contacted five weeks (± one week) after complete mobilization. All suspected venous thromboembolic events, including asymptomatic deep vein thrombosis, all deaths, and all bleeding events (with the exception of certain types of minor bleeding events defined in the protocol) will be reviewed by an independent adjudication committee blind to treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

* Requiring rigid or semi-rigid immobilization (e.g. with a plaster cast or brace) for at least 21 days and up to 45 days because of isolated non-surgical below-knee injury
* With a no weight-bearing recommendation at the time of inclusion (partial weight bearing is permitted e.g. crutches, walking cast, relief shoes),
* Presenting at least one of the following risk factors for venous thromboembolism: below-knee fracture or Achilles tendon rupture, age ≥40 years, body mass index > 30 kg/m2, oestrogen-containing hormonal replacement therapy or oral contraception, active cancer (treatment ongoing or stopped for less than one year), history of VTE, congenital or acquired hypercoagulable state,
* Requiring thromboprophylaxis according to the Investigator's judgement up to complete mobilization (corresponding to cast or brace removal)
* Able and willing to provide written informed consent

Exclusion Criteria:

* Delay between injury and randomization greater than two days,
* Treatment with antithrombotic or anticoagulant therapy, including low-dose anticoagulation, for more than 2 days prior to randomization,
* Anticoagulant therapy required or likely to be required during the study period for another reason (e.g. planned surgery justifying pharmacological thromboprophylaxis, curative dose for treatment of VTE, etc.)
* Known hypersensitivity to fondaparinux or nadroparin or their excipient,
* Known history of heparin-induced thrombocytopenia,
* Women of childbearing potential not using a reliable contraceptive method throughout the study period,
* Women pregnant or breast-feeding during the study period.
* Active, clinically significant bleeding,
* Clinically significant bleeding within the past six months,
* Major surgery within the previous three months,
* Intraocular (other than cataract), spinal, and/or brain surgery within the previous twelve months,
* Haemorrhagic stroke within the previous twelve months,
* Severe head injury within the previous three months,
* Documented congenital or acquired bleeding tendency/disorder(s),
* Previous (within 12 months) or active or currently treated peptic ulcer disease,
* Uncontrolled arterial hypertension (systolic blood pressure over 180 mm Hg or diastolic blood pressure over 110 mm Hg),
* Treatment with more than one antiplatelet agents (e.g. clopidogrel and aspirin) at any dose,
* Need for chronic aspirin at doses≥ 325 mg or chronic NSAIDs,
* Bacterial endocarditis,
* Severe hepatic impairment,
* Calculated creatinine clearance < 30 mL/min,
* Thrombocytopenia ( <100x10_9/L)
* Body weight < 50 kg.
* Any condition that could prevent the patient from providing written informed consent or from adhering to study treatment,
* Life expectancy under six months,
* Participation in any study using an investigational drug during the previous three months,
* Patient in whom V3 is unlikely to be feasible (e.g. patient moving house),
* In France, a subject will not be eligible for inclusion in this study if not either affiliated to or a beneficiary of a social security system. This is an additional exclusion criterion only applying to subjects enrolled in France.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1351 (Actual)
Dates: Start 2008-12; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (104):
- France (27):
  - GSK Investigational Site, Agen
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Antony
  - GSK Investigational Site, Argenteuil
  - GSK Investigational Site, Beauvais
  - GSK Investigational Site, Bobigny
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Cergy-Pontoise
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Colmar
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Mougins
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Orthez
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pringy
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Roanne
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Saint-Pierre
  - GSK Investigational Site, Sainte Colombe Les Vienne
  - GSK Investigational Site, Saintes
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Valenciennes
- Germany (15):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Gevelsberg, North Rhine-Westphalia
  - GSK Investigational Site, Moers, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Schmiedeberg, Saxony
  - GSK Investigational Site, Zwickau, Saxony
  - GSK Investigational Site, Zerbst, Saxony-Anhalt
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Altenburg, Thuringia
- Italy (12):
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Udine, Friuli Venezia Giulia
  - GSK Investigational Site, Latina, Lazio
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Bergamo, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Orbassano (TO), Piedmont
  - GSK Investigational Site, Catania, Sicily
  - GSK Investigational Site, Siena, Tuscany
  - GSK Investigational Site, Conegliano (TV), Veneto
  - GSK Investigational Site, Padua, Veneto
- Netherlands (6):
  - GSK Investigational Site, Amersfoort
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, Sittard-geleen
  - GSK Investigational Site, Utrecht
  - GSK Investigational Site, Venlo
- Russia (18):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Kursk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saint Petersburgh
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Stavropol
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Tver'
  - GSK Investigational Site, Tyumen
  - GSK Investigational Site, Ufa
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg
- Spain (26):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Aravaca
  - GSK Investigational Site, Avilés/Asturias
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Castellon
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Don Benito/Badajoz
  - GSK Investigational Site, Ferrol. La Coruña
  - GSK Investigational Site, Getafe/Madrid
  - GSK Investigational Site, Jaén
  - GSK Investigational Site, Linares
  - GSK Investigational Site, Lugo
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda/Madrid
  - GSK Investigational Site, Mondragón - Guipúzcoa
  - GSK Investigational Site, Ourense
  - GSK Investigational Site, Palencia
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Pozoblanco/Córdoba
  - GSK Investigational Site, San Sebastián de Los Reyes/Madrid
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Torrelodones/Madrid
  - GSK Investigational Site, Torrevieja
  - GSK Investigational Site, Valdemoro/Madrid
  - GSK Investigational Site, Vigo/Pontevedra

RESULTS

PARTICIPANT FLOW:
Groups:
- Nadroparin: 2850 anti-Xa International Units (IU) nadroparin calcium (in 0.3 milliliters [ml] in disposable prefilled syringes) was injected once daily subcutaneously after randomization (Day 1) until the end of immobilization and treatment period Day 45 (Visit 3)
- Fondaparinux: 2.5 milligrams (mg) fondaparinux sodium (in 0.5 ml) or 1.5 mg fondaparinux (in 0.3 ml) (in participants with creatinine clearance between 30 and 50 ml per minute) was injected once daily subcutaneously from Day 1 until Day 45 (Visit 3)
Period: Overall Study
Arm/Group | Nadroparin | Fondaparinux
Started | 622 | 621
Completed | 614 | 607
Not Completed | 8 | 14
Not completed — Adverse Event | 0 | 3
Not completed — Lost to Follow-up | 4 | 4
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Immobilization Stopped | 1 | 0
Not completed — Investigator/Orthopedic Surgeon Decision | 1 | 1
Not completed — Orthopedic Surgery | 0 | 2
Not completed — Visit Not Performed | 1 | 0
Not completed — Deep-vein Thrombosis | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nadroparin | Fondaparinux | Total
Number analyzed (Participants) | 622 | 621 | 1243
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristic data was collected in members of the Intent-to-Treat (ITT) Population, comprised of all randomized patients (recorded in the Interactive Voice Response System [IVRS] database) with a venous thromboembolism (VTE) status or experiencing death.
  Years
    Years | 46.5 (15.7) | 46.1 (16.0) | 46.3 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristic data was collected in members of the Intent-to-Treat (ITT) Population, comprised of all randomized patients (recorded in the Interactive Voice Response System [IVRS] database) with a venous thromboembolism (VTE) status or experiencing death.
  Participants
    Female | 336 | 328 | 664
    Male | 286 | 293 | 579

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Venous Thromboembolism (VTE) or Death up to the Time of Complete Mobilization
Description: VTE is defined as asymptomatic deep vein thrombosis (DVT: the formation of a blood clot in a deep vein) detected by systematic compression ultrasonography, symptomatic DVT, or symptomatic fatal or non-fatal pulmonary embolism (PE). An embolism is a clot in the blood that forms and blocks a blood vessel. A pulmonary embolism is a blood clot that has travelled from elsewhere in the body through the blood stream to block the main artery of the lung or one of its branches. All venous thromboembolic events and deaths were adjudicated by the independent Central Adjudication Committee (CAC).
Time Frame: Day 1 to complete mobilization plus 2 days (average of 35.9 study days)
Population: Intent-to-Treat (ITT) Population: all randomized participants with a VTE status or experiencing death. Participants without evaluation of the primary endpoint in the timeframe requested by the protocol were considered as missing data and therefore not included in the primary efficacy analysis.
Measure: Number; unit: participants
Arm/Group | Nadroparin | Fondaparinux
Number analyzed (Participants) | 586 | 584
participants | 48 | 15
Statistical Analysis 1: Comparison: Nadroparin vs Fondaparinux; Test type: Superiority or Other; p < 0.001, Fisher Exact; Odds Ratio (OR) = 0.30, 95% CI 2-sided [0.15 to 0.54]

2. Secondary Outcome: Number of Participants With Any Adjudicated Components of VTE, Asymptomatic DVT, Symptomatic DVT, Symptomatic PE, and Death
Description: All components of the primary endpoint were considered separately: any VTE; symptomatic (providing no evidence of disease existence) DVT (the formation of a blood clot in a deep vein) detected by systematic compression ultrasonography; symptomatic(providing evidence of disease existence) DVT; symptomatic PE (blood clot that has travelled from elsewhere in the body through the blood stream to block the main artery of the lung of one of its branches); and death.
Time Frame: Day 1 to complete mobilization plus 2 days (average of 35.7 study days)
Population: ITT Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Nadroparin | Fondaparinux
Number analyzed (Participants) | 622 | 621
participants
  Any VTE, n=586, 583 | 48 | 14
  Any asymptomatic DVT, n=585, 582 | 42 | 11
  Any symptomatic DVT, n=622, 621 | 7 | 2
  Any symptomatic PE, n=622, 621 | 0 | 2
  Death, n=622, 621 | 0 | 1

3. Secondary Outcome: Number of Participants With Confirmed VTE and Death up to the Final Visit or Contact
Description: The number of participants with VTE (defined as asymptomatic deep vein thrombosis [DVT: the formation of a blood clot in a deep vein] detected by systematic compression ultrasonography, symptomatic DVT, or symptomatic fatal or non-fatal pulmonary embolism [PE]) and death was assessed. An embolism is a clot in the blood that forms and blocks a blood vessel. A PE is a blood clot that has travelled from elsewhere in the body through the blood stream to block the main artery of the lung or one of its branches.
Time Frame: Day 1 to 5 weeks (plus or minus 1 week) after complete mobilization (average of 67.8 study days)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Nadroparin | Fondaparinux
Number analyzed (Participants) | 622 | 621
participants | 49 | 15

4. Secondary Outcome: Number of Participants With Major Bleeding From Day 1 to Complete Mobilization and From Day 1 up to the Final Visit or Contact
Description: Major bleeding is defined as bleeding that results in a fatality, symptomatic bleeding in a critical area or organ, bleeding causing a fall in hemoglobin level of 20 grams/liter (1.24 millimoles/liter) or more compared with the pre-randomization hemoglobin level, or bleeding that leads to a transfusion of two or more units of whole blood or red blood cells. All episodes of bleeding were adjudicated by an independent CAC. The committee members were unaware of the participants' treatment assignment.
Time Frame: Day 1 to complete mobilization plus 4 days (average of 37.7 study days); Day 1 up to final visit or contact (average of 66.3 study days)
Population: As-Treated Population: all participants who received at least one dose of study treatment
Measure: Number; unit: participants
Arm/Group | Nadroparin | Fondaparinux
Number analyzed (Participants) | 670 | 674
participants
  Up to complete mobilization plus 4 days | 0 | 1
  Up to the final visit or contact | 0 | 1

5. Secondary Outcome: Number of Participants With Clinically Relevant Non-major Bleeding From Day 1 to Complete Mobilization and From Day 1 up to the Final Visit or Contact
Description: Clinically relevant non-major bleeding that does not qualify as major is defined as bleeding leading to treatment discontinuation, and/or epistaxis (bleeding through the nose) that lasts for more than 5 minutes or necessitates intervention (e.g., packing), spontaneous macroscopic haematuria (blood in urine), gastrointestinal haemorrhage, haemoptysis (coughing up blood), or subcutaneous haematoma (localized collection of blood) > 100 centimeters squared. All episodes of bleeding were adjudicated by an independent CAC. The committee members were unaware of the participants' treatment assignment.
Time Frame: as for outcome 4
Population: As-Treated Population
Measure: Number; unit: participants
Arm/Group | Nadroparin | Fondaparinux
Number analyzed (Participants) | 670 | 674
participants
  Up to complete mobilization plus 4 days | 3 | 1
  Up to the final visit or contact | 4 | 1

6. Secondary Outcome: Number of Participants With Minor Bleeding From Day 1 to Complete Mobilization and From Day 1 up to the Final Visit or Contact
Description: Minor bleeding is defined as clinically overt bleeding events that do not meet the criteria for major or clinically relevant non-major bleeding. All episodes of bleeding were adjudicated by an independent CAC. The committee members were unaware of the participants' treatment assignment.
Time Frame: as for outcome 4
Population: As-Treated Population
Measure: Number; unit: participants
Arm/Group | Nadroparin | Fondaparinux
Number analyzed (Participants) | 670 | 674
participants
  Up to complete mobilization plus 4 days | 3 | 9
  Up to the final visit or contact | 3 | 9

7. Secondary Outcome: Participants With Any Incidence of Any Bleeding Event as Adjudicated by a CAC) From Day 1 to Complete Mobilization and From Day 1 up to the Final Visit or Contact
Description: All episodes of bleeding, except minor bruising, skin hematomas not greater than 5 centimeters in diameter, self-limited epistaxis (bleeding through the nose), and self-limited gingival (gum) bleeding, were adjudicated by an independent CAC. The committee members were unaware of the participants' treatment assignment.
Time Frame: as for outcome 4
Population: As-Treated Population
Measure: Number; unit: participants
Arm/Group | Nadroparin | Fondaparinux
Number analyzed (Participants) | 670 | 674
participants
  Up to complete mobilization plus 4 days | 6 | 11
  Up to the final visit or contact | 7 | 11

ADVERSE EVENTS:
Description: Serious adverse events (SAEs) and non-serious AEs were collected in members of the As-Treated Population, comprised of all participants having received at least one dose of study treatment.
Arm/Group | Nadroparin | Fondaparinux
Serious Adverse Events (participants affected / at risk) | 9/670 | 6/674
Other Adverse Events (participants affected / at risk) | 95/670 | 93/674
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nadroparin (N=670) | Fondaparinux (N=674)
Appendicitis (Infections and infestations) | 0 | 1
Haematoma infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0
Fracture malunion (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nadroparin (N=670) | Fondaparinux (N=674)
Headache (Nervous system disorders) | 33 | 24
Injection site haematoma (General disorders) | 31 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 21
Nausea (Gastrointestinal disorders) | 10 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 14
Lymphadenopathy (Blood and lymphatic system disorders) | 13 | 8
Oedema peripheral (General disorders) | 7 | 11
Dizziness (Nervous system disorders) | 6 | 7
Hypertension (Vascular disorders) | 8 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 6
Haematoma (Vascular disorders) | 1 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.